CLINICAL TRIAL: NCT02893683
Title: Paris Visual Learning Test (PVLT): a New French Task for Assess Visual Learning and Memory to Multiple Sclerosis Patients
Brief Title: Paris Visual Learning Test: a New French Task for Assess Visual Learning and Memory to Multiple Sclerosis Patients
Acronym: valid-PVLT
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: OGT_2013-4
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis
Keywords: Paris Visual Learning Test; visual memory; criterion validity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

INTERVENTIONS:
Other: Paris Visual Learning Test

SUMMARY:
Cognitive impairment affects up to 65% of multiple sclerosis (MS) subjects, especially memory function.

Rothschild Foundation has developped the Paris Visual Learning and memory Test (PVLT). 165 healthy volunteers were studied for its normalization.

The main objective of the present study is to assess the validity of PVLT by comparing MS patients' test results to a database including the test results of 280 healthy control subjects, following recommended international standards.

ELIGIBILITY:
Inclusion Criteria:

* multiple sclerosis
* 20-89 years old

Exclusion Criteria:

* acute inflammatory stage of central nervous system (< 1 month)
* other neurological or psychiatric disease
* regular drug and/or alcohol consumption
* refusal to participate in the study
* no health insurance coverage
* patient under legal protection

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis. The test results will be compared to a database including results of healthy control patients.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
test score | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire VIRET-VILAYPHONH, Study Director — Fondation OPH A de Rothschild; Olivier GOUT, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France